CLINICAL TRIAL: NCT02709577
Title: A Pilot Feasibility Sham Controlled Study of the GI Sleeve for the Treatment of Type 2 Diabetes
Brief Title: A Study of the GI Sleeve for the Treatment of Type 2 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Morphic Medical Inc. (Industry)
Collaborators: Hospital Dipreca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-5
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- EndoBarrier Gastrointestinal Liner (Experimental): Subjects randomized and implanted with the EndoBarrier Gastrointestinal liner; subjects will be implanted for 24 weeks to 52 weeks and evaluated for study endpoints.
  Interventions: Device: EndoBarrier Gastrointestinal Liner
- Sham: endoscopy and standard of care (Experimental): Subjects randomized to sham arm received an upper GI examination and were evaluated for study endpoints.
  Interventions: Other: Sham: endoscopy and standard of care

INTERVENTIONS:
Device: EndoBarrier Gastrointestinal Liner — The EndoBarrier is a single use, implant consisting of a tube of composite material which is placed in the proximal section of the duodenum. The implant is fixed in place with the aid of a metal anchor. The device is delivered via an endoscope. The implant facilitates the passage of food from the stomach through the tube to the proximal section of the jejunum.
  Other Names: GI Sleeve
  Arms: EndoBarrier Gastrointestinal Liner
Other: Sham: endoscopy and standard of care — Sham subjects had an endoscopic procedure and then received standard of care treatment of their diabetes
  Other Names: Control
  Arms: Sham: endoscopy and standard of care

SUMMARY:
The purpose of the study was to evaluate the safety and efficacy of the EndoBarrier Gastrointestinal Liner compared to sham control in subjects with Type 2 diabetes.

DETAILED DESCRIPTION:
The study was designed as a randomized, single blind, sham controlled, pilot efficacy study of subjects with Type 2 diabetes enrolled at 2 centers in Santiago, Chile. Subjects were enrolled at a 2:1 ratio (EndoBarrier to sham). Following implantation or sham procedure, subjects were treated for 24 weeks or 52 weeks. Following explant, subjects were followed for an additional 8-12 weeks.

Subject evaluations included measurements of HbA1c, glucose, insulin, weight, changes in diabetic medications, and meal tolerance tests. Safety was monitored through the collection of clinical labs, physical assessments, endoscopy and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 55 years - Male or Female
* Patients with type 2 diabetes, treated for 10 years or less
* HbA1c level ≥ 7.0 and ≤ 10.0%
* Fasting glucose ≤ 240 mg/dl
* Patients taking metformin, sulfonylureas or thiazolidinediones (TZDs), either alone or in combination
* BMI > 30 and <50
* Patients willing to comply with study requirements
* Patients who have signed an informed consent form
* Women who are post-menopausal, surgically sterile, or on oral contraceptives for at least three months and who do not plan on becoming pregnant during the course of the study.

Exclusion Criteria:

* Patients taking oral medications to control their diabetes other than sulfonylureas, metformin or thiazolidinediones
* Patients diagnosed with type 1 diabetes mellitus or had a history of ketoacidosis
* Patients requiring insulin
* Patients with lab evidence of probable insulin production failure (fasting C peptide serum level < 1ng/ml)
* Patients with a weight loss of > 10 lbs within the three months of screening
* Patients requiring prescription anticoagulation therapy
* Patients with iron deficiency and iron deficiency anemia
* Patients with a history of abnormal pathologies of the GI tract
* Patients with known gallstones or kidney stones prior to implant
* Known infection at the time of implant
* Severe coagulopathy, upper gastro-intestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasia
* Pregnant or has the intention of becoming pregnant in the next 12 months
* Patients with a history of active kidney stones
* Mentally retarded or emotionally unstable, or exhibits psychological characteristics which, in the opinion of the investigator, makes the subject a poor candidate for device placement or clinical trial
* Previous GI surgery that could affect the ability to place the sleeve or the function of the implant
* Patients unable to discontinue NSAIDs (non-steroidal anti-inflammatory drugs) during the implant period
* H. pylori positive patients (Note: patients may be enrolled if they had a prior history and were successfully treated)
* Patients receiving weight loss medications such as Meridia and Xenical
* Family or patient history of a known diagnosis or pre-existing symptom of systemic lupus erythematous, scleroderma or other autoimmune connective tissue disorder
* Patients with Gastrointestinal Reflux Disease (GERD)
* Participating in another ongoing investigational clinical trial
* Patients taking corticosteroids or drugs known to affect gastrointestinal motility (such as reglan)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Rodriguez Grunert, MD, Principal Investigator — Hospital Dipreca

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: EndoBarrier Gastrointestinal Liner: Subjects in Cohort A were implanted with the device for 24 weeks and given the option to continue for up to 52 weeks.
- Cohort B:EndoBarrier Gastrointestinal Liner: Subjects in Cohort B had a 52 week implant period. Follow-up after device removal was originally 6 months and then extended to 12 months based on physician discretion.
- Cohort A Control Sham: Device was not implanted
- Cohort B Control Sham: Device not implanted.
Period: Overall Study
Arm/Group | Cohort A: EndoBarrier Gastrointestinal Liner | Cohort B:EndoBarrier Gastrointestinal Liner | Cohort A Control Sham | Cohort B Control Sham
Started | 12 | 13 | 6 | 5
Completed | 10 | 8 | 4 | 5
Not Completed | 2 | 5 | 2 | 0
Not completed — non-accommodating anatomy | 0 | 1 | 0 | 0
Not completed — procedural complication | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Device Cohort A had 10 Subjects, Device Cohort B had 8 subjects, Sham Cohort A had 4 subjects and Sham Cohort B had 5 subjects at Baseline
Groups:
- Total: Total of all reporting groups
Arm/Group | EndoBarrier Gastrointestinal Liner | Sham: Endoscopy and Standard of Care | Total
Number analyzed (Participants) | 18 | 9 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] — Cohort A and Cohort B
  years
    Cohort A | 44.8 (7.96) | 52.1 (16.14) | 46.9 (10.75)
    Cohort B | 41.2 (9.28) | 46.3 (6.25) | 46.1 (8.36)
Gender [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  Chile | 18 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c Values From Baseline Measurement
Description: Cohort A: Assessment of improvement in the glycemic control defined as a change in HbA1c values from baseline.
  Cohort B. Assessment of improvement in glycemic control defined as a change in HbA1c values of at least 0.5% from baseline.
Time Frame: Baseline to 24 weeks or 52 weeks
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Groups:
- Cohort B: EndoBarrier Gastrointestinal Liner: Subjects in Cohort B had a 52 week implant period. Follow-up after device removal was originally 6 months and then extended to 12 months based on physician discretion.
- Cohort A Control Sham: Endoscopy and Standard of Care; Cohort B Control Sham: Endoscopy and Standard of Care: Subjects received only an upper GI endoscopic examination with no device implantation.
Arm/Group | Cohort A: EndoBarrier Gastrointestinal Liner | Cohort B: EndoBarrier Gastrointestinal Liner | Cohort A Control Sham: Endoscopy and Standard of Care | Cohort B Control Sham: Endoscopy and Standard of Care
Number analyzed (Participants) | 10 | 8 | 4 | 5
percentage of HbA1c | 2.4 (1.96) | 2.2 (1.44) | 0.8 (0.81) | 1.6 (1.05)

2. Secondary Outcome: Absolute Weight Change
Time Frame: 24 weeks or 52 weeks
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Cohoart A: EndoBarrier Gastrointestinal Liner: Subjects in Cohort A were implanted with the device for 24 weeks and given the option to continue for up to 52 weeks.
- Cohort A Control Sham: Endoscopy and Standard of Care: Subjects received only an upper GI endoscopic examination with no device implantation. Follow-up after treatment phase was originally 6 months and then extended to 12 months based on physician discretion.
- Cohort B Control Sham: Endoscopy and Standard of Care: Subjects received only an upper GI endoscopic examination with no device implantation. Follow-up after treatment phase was 12 months.
Arm/Group | Cohoart A: EndoBarrier Gastrointestinal Liner | Cohort B: EndoBarrier Gastrointestinal Liner | Cohort A Control Sham: Endoscopy and Standard of Care | Cohort B Control Sham: Endoscopy and Standard of Care
Number analyzed (Participants) | 10 | 8 | 4 | 5
kg | 9.9 (1.7) | 11.3 (2.0) | 7.9 (5.4) | 5.4 (3.7)

ADVERSE EVENTS:
Time Frame: I year
Groups:
- Cohorts A and B: EndoBarrier Gastrointestinal Liner: Subjects randomized and implanted with the EndoBarrier Gastrointestinal liner; subjects will be implanted for 24 or 52 weeks and evaluated for study endpoints
- Cohorts A and B Sham: Endoscopy and Standard of Care: Subjects randomized to sham and underwent an endoscopy procedure and then received standard of care treatment for their diabetes
Arm/Group | Cohorts A and B: EndoBarrier Gastrointestinal Liner | Cohorts A and B Sham: Endoscopy and Standard of Care
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/11
Other Adverse Events (participants affected / at risk) | 25/25 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohorts A and B: EndoBarrier Gastrointestinal Liner (N=25) | Cohorts A and B Sham: Endoscopy and Standard of Care (N=11)
Oesophageal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohorts A and B: EndoBarrier Gastrointestinal Liner (N=25) | Cohorts A and B Sham: Endoscopy and Standard of Care (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 10 (10) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 25 (51) | 8 (8)
Constipation (Gastrointestinal disorders) | 7 (7) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 2 (2)
Erosive duodenitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (11) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 17 (17) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Folliculitis (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 4 (4) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 7 (7) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 7 (7) | 0 (0)
Blood cholesterol increased (Investigations) | 2 (2) | 0 (0)
Blood iron decreased (Investigations) | 4 (4) | 0 (0)
High density lipoprotein decreased (Investigations) | 1 (1) | 0 (0)
Low density lipoprotein decreased (Investigations) | 1 (1) | 0 (0)
Serum ferritin decreased (Investigations) | 2 (2) | 0 (0)
ECG signs of myocardial ischaemia (Investigations) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 23 (23) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 7 (7) | 7 (7)
Anxiety disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 5 (5) | 4 (4)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less